CLINICAL TRIAL: NCT00380692
Title: A Randomized, Double-blind Comparison of Atomoxetine Hydrochloride and Placebo for Symptoms of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents With Autism Spectrum Disorder
Brief Title: Atomoxetine Versus Placebo for Symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in Children and Adolescents With Autism Spectrum Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10483; B4Z-UT-S017 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Autistic Disorder; Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Atomoxetine (Experimental): atomoxetine 0.5 mg/kg/day every day (QD), by mouth (PO) for 1 week, atomoxetine 0.8mg/kg/day QD, PO for 1 week, 1.2mg/kg/day QD, PO for 6 weeks then atomoxetine 0.5-1.2 mg/kg/day QD, PO for up to 20 weeks
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): placebo every day (QD), by mouth (PO) for 8 weeks
  Then patients can take atomoxetine 0.5-1.2 mg/kg/day QD, PO up to 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine
  Other Names: LY139603; Strattera
  Arms: Atomoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether atomoxetine is effective in reducing ADHD (Attention Deficit/Hyperactivity Disorder) symptoms in children and adolescents with ASD (Autism Spectrum Disorder).

ELIGIBILITY:
Inclusion Criteria (most important):

* ASD (autistic disorder or Asperger's disorder or Pervasive Developmental Disorder - Not Otherwise Specified [PDD NOS])
* Criteria A through D for Attention-Deficit/Hyperactivity Disorder (ADHD)
* At least 1.5 standard deviations above the age norm for their diagnostic subtype using published norms for the ADHD Rating Scale-IV-Parent Version
* Intelligence quotient (IQ) score > 60

Exclusion Criteria (most important):

* weight under 20 kg
* Patients who meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) criteria for ASD other than Autistic Disorder, PDD-NOS or Asperger's Disorder;history of Bipolar I or II disorder, schizophrenia, another psychotic disorder, substance abuse;Have a significant medical condition such as heart disease, hypertension, liver or renal failure, pulmonary disease, or seizure disorder identified by history, physical examination, or laboratory tests; Patients who have taken (or are currently taking) anticonvulsants for seizure control.
* patients at serious suicidal risk.
* Contraindication to the use of atomoxetine
* Patients who in the investigator's judgment are likely to need psychotropic medications apart from the drug. Patients who at any time during Study Period II are likely to begin a structured psychotherapy, likely to require hospitalization (i.e. in-patient treatment) or likely to be dismissed from in-patient treatment. Psychotherapy (including hospitalization) initiated at least 2 months prior to study participation is acceptable; however, after study participation has begun, only during Study Period III supportive or educational therapy is permitted.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- Netherlands (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoorn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oosterhout
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Hague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Utrecht

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Harfterkamp M, Buitelaar JK, Minderaa RB, van de Loo-Neus G, van der Gaag RJ, Hoekstra PJ. Atomoxetine in autism spectrum disorder: no effects on social functioning; some beneficial effects on stereotyped behaviors, inappropriate speech, and fear of change. J Child Adolesc Psychopharmacol. 2014 Nov;24(9):481-5. doi: 10.1089/cap.2014.0026. Epub 2014 Nov 4. PMID 25369243
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] van der Meer JM, Harfterkamp M, van de Loo-Neus G, Althaus M, de Ruiter SW, Donders AR, de Sonneville LM, Buitelaar JK, Hoekstra PJ, Rommelse NN. A randomized, double-blind comparison of atomoxetine and placebo on response inhibition and interference control in children and adolescents with autism spectrum disorder and comorbid attention-deficit/hyperactivity disorder symptoms. J Clin Psychopharmacol. 2013 Dec;33(6):824-7. doi: 10.1097/JCP.0b013e31829c764f. No abstract available. PMID 24018545
- [Derived] Harfterkamp M, Buitelaar JK, Minderaa RB, van de Loo-Neus G, van der Gaag RJ, Hoekstra PJ. Long-term treatment with atomoxetine for attention-deficit/hyperactivity disorder symptoms in children and adolescents with autism spectrum disorder: an open-label extension study. J Child Adolesc Psychopharmacol. 2013 Apr;23(3):194-9. doi: 10.1089/cap.2012.0012. Epub 2013 Apr 11. PMID 23578015
- [Derived] Harfterkamp M, van de Loo-Neus G, Minderaa RB, van der Gaag RJ, Escobar R, Schacht A, Pamulapati S, Buitelaar JK, Hoekstra PJ. A randomized double-blind study of atomoxetine versus placebo for attention-deficit/hyperactivity disorder symptoms in children with autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2012 Jul;51(7):733-41. doi: 10.1016/j.jaac.2012.04.011. Epub 2012 May 25. PMID 22721596
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I was a screening and wash-out period. Study Period II (visits 2-6) was an 8-week double-blind period. Patients were randomized at Visit 2. Study Period III (visits 6-11) was a 20-week open-label extension period. Treatment groups in Study Period III refer to treatment group assignment during Double-Blind Period.
Groups:
- Atomoxetine: atomoxetine: 0.5 mg/kg/day daily (QD), by mouth (PO) for 1 week, atomoxetine 0.8mg/kg/day QD, PO for 1 week, 1.2mg/kg/day QD, PO for 6 weeks then atomoxetine 0.5-1.2 mg/kg/day QD, PO for up to 20 weeks.
- Placebo: placebo: daily (QD), by mouth (PO) for 8 weeks.
  Then patients can take atomoxetine 0.5-1.2 mg/kg/day QD, PO up to 20 weeks.
Period: Study Period II - Double Blind
Arm/Group | Atomoxetine | Placebo
Started | 48 | 49
Completed | 43 | 46
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Parent/Caregiver Decision | 1 | 0
Period: Study Period III - Open Label
Arm/Group | Atomoxetine | Placebo
Started | 42 (One patient who completed Study Period II did not enter Study Period III.) | 46
Completed | 36 | 34
Not Completed | 6 | 12
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Lack of Efficacy | 0 | 4
Not completed — Parent/Caregiver Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 48 | 49 | 97
Age Continuous [Mean (Standard Deviation); unit: years] | 9.9 (2.72) | 10.0 (2.90) | 9.9 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 42 | 41 | 83
Region of Enrollment [Number; unit: participants]
  Netherlands | 48 | 49 | 97
Race/Ethnicity [Number; unit: participants]
  Caucasian | 48 | 47 | 95
  African | 0 | 1 | 1
  Hispanic | 0 | 1 | 1
Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version- Total Score [Mean (Standard Deviation); unit: units on a scale] — Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders, Version IV (DSM-IV) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
  units on a scale | 40.7 (7.47) | 38.6 (8.43) | 39.6 (8.00)
Autism Diagnostic Interview-Revised (ADI-R) [Mean (Standard Deviation); unit: units on a scale] — ADI-R is a highly structured method of eliciting information from a parent to confirm clinical impression of autism. To meet criteria for autism, child must meet criteria in each of 3 content areas (communication [cutoff score=8 for verbal, 7 for nonverbal], social interaction [cutoff score=10], restricted/repetitive behavior [cutoff score=3]).
  units on a scale | 37.4 (12.45) | 37.2 (9.68) | 37.3 (11.09)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter squared] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilogram/meter squared | 18.5 (3.40) | 18.1 (3.36) | 18.3 (3.37)
Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale [Mean (Standard Deviation); unit: units on a scale] — Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
  units on a scale | 5.0 (0.74) | 5.1 (0.90) | 5.1 (0.83)
Height [Mean (Standard Deviation); unit: centimeters] | 146.0 (16.57) | 148.0 (19.11) | 147.0 (17.84)
Score for Performance IQ [Mean (Standard Deviation); unit: units on a scale] — Performance IQ was assessed with the Wechsler Intelligence Scales (WISC-III). There are 5 performal subtests consisting of nonverbal problems, all of which are timed and some of which allow bonus points for extra fast work. The mean score is 100.
  units on a scale | 89.9 (16.59) | 94.9 (17.46) | 92.4 (17.14)
Score for Verbal IQ [Mean (Standard Deviation); unit: units on a scale] — Verbal IQ was assessed with the Wechsler Intelligence Scales (WISC-III). There are 5 verbal subtests consisting of oral questions without time limits except for Arithmetic. The mean score is 100.
  units on a scale | 93.2 (18.49) | 94.4 (18.26) | 93.8 (18.29)
Score for the Overall Scale Intelligence [Mean (Standard Deviation); unit: units on a scale] — Overall scale intelligence was assessed with the Wechsler Intelligence Scales (WISC-III). The mean score is 100.
  units on a scale | 91.0 (16.41) | 94.6 (17.71) | 92.9 (17.08)
Weight [Mean (Standard Deviation); unit: kilograms] | 41.0 (14.92) | 41.5 (16.12) | 41.2 (15.46)

OUTCOME MEASURES:

1. Primary Outcome: ADHD Rating Scale-IV-Parent Version: Investigator Scored - Total Score
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders, Version IV (DSM-IV) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
Time Frame: Baseline and 8 weeks
Population: Number of randomized participants with a value at baseline and 8 week endpoint. Last Observation Carried Forward analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
units on a scale
  Baseline Total Score (n=48, n=49) | 40.7 (7.47) | 38.6 (8.43)
  8 Week Endpoint Total Score (n=43, n=47) | 32.3 (10.97) | 37.3 (9.57)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for treatment group differences over time; Mean Difference (Net) = -6.7, 95% CI [-10.0 to -3.4], Standard Error of Mean 1.7

2. Secondary Outcome: Clinical Global Impressions-ADHD-Improvement (CGI-ADHD - I)
Description: Measures total improvement (or worsening) of a patient's ADHD symptoms from the beginning of treatment (1=very much improved, 7=very much worsened).
Time Frame: 8 weeks, 28 weeks
Population: Number of randomized participants with values at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 43 | 46
units on a scale
  8 Week Improvement Score | 3.5 (1.08) | 3.9 (0.96)
  28 Week Improvement Score (n=39, n=35) | 2.5 (1.14) | 2.7 (1.05)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.921, Mixed Models Analysis — P-value for treatment differences over time; Mean Difference (Net) = -0.0, 95% CI [-0.5 to 0.4], Standard Error of Mean 0.2

3. Secondary Outcome: Conners' Teacher Rating Scale - Revised: Short Form (CTRS-R:S)
Description: A 28-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the teacher to assess problem behaviors related to ADHD. Subscale total scores range from 0 to 15 for Oppositional and Cognitive Problems, 0 to 21 for Hyperactivity, and 0 to 36 for ADHD Index.
Time Frame: Baseline, 8 weeks, 28 weeks
Population: Number of randomized participants who had a value at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 42 | 44
units on a scale
  Oppositional: Baseline (n=42, n=44) | 4.1 (3.54) | 3.6 (3.53)
  Oppositional: 8 Week (n=36, n=36) | 3.8 (4.43) | 3.4 (3.35)
  Oppositional: 28 Week (n=26, n= 25) | 2.3 (3.33) | 1.4 (1.98)
  Hyperactivity: Baseline (n=42, n=44) | 8.8 (5.50) | 8.2 (5.06)
  Hyperactivity: 8 Week (n=36, n=36) | 7.6 (5.54) | 8.3 (5.63)
  Hyperactivity: 28 Week (n=26, n=25) | 6.0 (4.90) | 5.2 (4.13)
  Cognitive/Attention: Baseline (n=40, n=44) | 6.8 (4.45) | 4.8 (3.68)
  Cognitive/Attention: 8 Week (n=34, n=36) | 6.1 (4.56) | 4.6 (3.53)
  Cognitive/Attention: 28 Week (n=26, n=25) | 4.7 (3.58) | 4.6 (3.85)
  ADHD: Baseline (n=42, n=44) | 18.5 (9.27) | 18.1 (7.49)
  ADHD: 8 Week (n=36, n=36) | 15.8 (9.85) | 17.2 (8.69)
  ADHD: 28 Week (n=26, n=25) | 13.5 (8.61) | 12.5 (5.95)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.369, ANCOVA — P-value for treatment differences in Oppositional Score at 8 weeks; Mean Difference (Net) = -0.6, 95% CI [-1.8 to 0.7], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.024, ANCOVA — P-value for treatment differences in Hyperactivity score at 8 weeks; Mean Difference (Net) = -2.0, 95% CI [-3.7 to -0.3], Standard Error of Mean 0.87
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.179, ANCOVA — P-value for treatment differences in Cognititve/Attention score at 8 weeks; Mean Difference (Net) = -0.7, 95% CI [-1.7 to 0.3], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.077, ANCOVA — P-value for treatment differences in ADHD score at 8 weeks; Mean Difference (Net) = -2.7, 95% CI [-5.6 to 0.3], Standard Error of Mean 1.48

4. Secondary Outcome: ADHD Rating Scale-IV-Parent Version: Investigator Scored Total Score
Description: Measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
Time Frame: 28 weeks
Population: Randomized participants with a value at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 38 | 35
units on a scale | 23.6 (11.81) | 25.9 (10.58)

5. Secondary Outcome: Sleep Measure Scale
Description: 10-item parent-based scale assessing sleep problems (6 point Likert scale). Scores: Difficulty falling asleep (1-6); Quality of sleep (3-18); Functional outcome (6-36). Lower scores indicate higher problems with item. Open-ended items: Time to fall asleep (1 [0-15 minutes] to 5 [>1 hour]); Total hours (numbers associated with hours of sleep).
Time Frame: Baseline, 8 weeks, 28 weeks
Population: Randomized participants with a value at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
units on a scale
  Time to Fall Asleep: Baseline (n=48, n=49) | 2.9 (1.49) | 2.8 (1.41)
  Time to Fall Asleep: 8 Week (n=43, n=46) | 2.6 (1.43) | 3.0 (1.34)
  Time to Fall Asleep: 28 Week (n=35, n=35) | 3.1 (1.49) | 2.6 (1.14)
  Difficulty Falling Asleep: Baseline (n=48, n=49) | 3.4 (1.91) | 3.3 (1.58)
  Difficulty Falling Asleep: 8 Week (n=43, n=46) | 3.6 (1.80) | 3.3 (1.64)
  Difficulty Falling Asleep: 28 Week (n=38, n=36) | 3.2 (1.76) | 3.7 (1.69)
  Total Hours of Sleep: Baseline (n=48, n=49) | 9.1 (1.38) | 9.3 (1.46)
  Total Hours of Sleep: 8 Weeks (n=42, n=46) | 8.9 (1.49) | 9.1 (1.51)
  Total Hours of Sleep: 28 Week (n=36, n=34) | 8.9 (1.61) | 9.2 (1.12)
  Quality of Sleep: Baseline (n=48, n=49) | 14.1 (2.85) | 14.4 (2.84)
  Quality of Sleep: 8 Week (n=43, n=46) | 14.2 (3.08) | 14.9 (2.86)
  Quality of Sleep: 28 Week (n=38, n=36) | 14.6 (2.88) | 15.0 (2.35)
  Functional Outcome During Day:Baseline (n=48,n=49) | 29.6 (4.69) | 30.0 (4.07)
  Functional Outcome During Day:8 Week (n=43,n=46) | 29.1 (5.09) | 30.0 (4.80)
  Functional Outcome During Day:28Week (n=38,n=36) | 27.8 (6.38) | 29.6 (4.76)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.028, ANCOVA — P-value for treatment differences in Time to fall asleep score at 8 weeks; Mean Difference (Net) = -0.5, 95% CI [-1.0 to -0.1], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.407, ANCOVA — P-value for treatment differences in Difficulty falling asleep score at 8 weeks; Mean Difference (Net) = 0.3, 95% CI [-0.3 to 0.9], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.652, ANCOVA — P-value for treatment differences in Total hours of sleep score at 8 weeks; Mean Difference (Net) = -0.1, 95% CI [-0.6 to 0.4], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.112, ANCOVA — P-value for treatment differences in Quality of sleep score at 8 weeks; Mean Difference (Net) = -0.8, 95% CI [-1.7 to 0.2], Standard Error of Mean 0.49
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.188, ANCOVA — P-value for treatment differences in Functional outcome during day score at 8 weeks; Mean Difference (Net) = -1.1, 95% CI [-2.9 to 0.6], Standard Error of Mean 0.87

6. Secondary Outcome: Aberrant Behavior Checklist (ABC)
Description: The ABC is a 58-item informant-based scale comprised of five subscales (Irritability [15 items], Lethargy [16], Stereotypic Behaviors [7], Hyperactivity [16], Inappropriate Speech [4]). Individual item scores range from 0 (no problem) to 3 (severe problem). Subscale scores are total of individual item scores in subscale: Irritability (0-45); Lethargy (0-48); Stereotypic (0-21); Hyperactivity (0-48); Inappropriate Speech (0-12).
Time Frame: Baseline, 8 weeks, 28 weeks
Population: Randomized participants with values at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
units on a scale
  Irritiability: Baseline (n=47, n=49) | 17.4 (9.15) | 16.2 (9.49)
  Irritiability: 8 Week (n=43, n=46) | 14.5 (9.36) | 15.4 (9.80)
  Irritiability: 28 Week (n=38, n=36) | 11.5 (10.12) | 10.4 (8.05)
  Lethargy: Baseline (n=47, n=49) | 12.7 (8.33) | 12.5 (8.03)
  Lethargy: 8 Week (n=43, n=46) | 11.1 (9.34) | 11.5 (8.17)
  Lethargy: 28 Week (n=38 , n=36) | 7.5 (7.24) | 8.4 (6.64)
  Stereotypic: Baseline (n=47, n=49) | 6.6 (5.07) | 4.1 (4.47)
  Stereotypic: 8 Week (n=43, n=46) | 3.6 (4.01) | 3.6 (4.12)
  Stereotypic: 28 Week (n=38, n=36) | 3.3 (4.03) | 1.7 (2.77)
  Hyperactivity: Baseline (n=47, n=49) | 28.2 (9.40) | 25.5 (11.56)
  Hyperactivity: 8 Week (n=43, n=45) | 22.5 (11.05) | 24.6 (10.33)
  Hyperactivity: 28 Week (n=38, n=36) | 16.4 (12.17) | 16.0 (9.60)
  Inappropriate Speech: Baseline (n=47, n=49) | 4.8 (3.21) | 4.6 (3.35)
  Inappropriate Speech: 8 Week (n=43, n=46) | 3.8 (2.92) | 4.5 (3.26)
  Inappropriate Speech: 28 Week (n=38, n=36) | 3.1 (3.22) | 2.9 (2.35)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.452, ANCOVA — P-value for treatment differences in Irritability score at 8 weeks; Mean Difference (Net) = -1.0, 95% CI [-3.5 to 1.6], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.850, ANCOVA — P-value for treatment differences in Lethargy score at 8 weeks; Mean Difference (Net) = -0.2, 95% CI [-2.4 to 2.0], Standard Error of Mean 1.10
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.014, ANCOVA — P-value for treatment differences in Stereotypic score at 8 weeks; Mean Difference (Net) = -1.6, 95% CI [-2.8 to -0.3], Standard Error of Mean 0.63
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value for treatment differences in Hyperactivity score at 8 weeks; Mean Difference (Net) = -4.4, 95% CI [-7.8 to -1.1], Standard Error of Mean 1.68
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.045, ANCOVA — P-value for treatment differences in Inappropriate speech score at 8 weeks; Mean Difference (Net) = -0.9, 95% CI [-1.7 to -0.0], Standard Error of Mean 0.42

7. Secondary Outcome: Children's Social Behavior Questionnaire (CSBQ) Total Score
Description: CSBQ is filled out by parents and consists of 49 items. Items are rated in an ordinal rather than a discrete fashion in order to establish the extent to which problems are present. The CSBQ consists of six subscales. Individual item scores range from 0=does not apply to 2=applies clearly. Total score ranges from 0 to 98.
Time Frame: Baseline, 8 weeks, 28 weeks
Population: Randomized participants with value at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
units on a scale
  Baseline (n=48, n=49) | 53.6 (14.81) | 52.4 (15.97)
  8 Week (n=43, n=46) | 46.1 (15.88) | 50.2 (14.62)
  28 Week (n=38, n=35) | 40.4 (19.55) | 43.6 (17.26)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.069, ANCOVA — P-value for treatment differences in Total score at 8 weeks; Mean Difference (Net) = -3.9, 95% CI [-8.1 to 0.3], Standard Error of Mean 2.13

8. Secondary Outcome: General Health Questionnaire (GHQ) Total Score
Description: Parental distress is measured with the GHQ. The raw total score (based on 0-0-1-1 scoring system) can be used as an overall index of psychological distress, ranging from 0 to 12 with higher scores indicating more distress.
Time Frame: Baseline, 8 weeks, 28 weeks
Population: Randomized participants with value at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
units on a scale
  Baseline (n=48, n=49) | 2.9 (3.45) | 4.0 (3.79)
  8 Week (n=43, n=46) | 2.3 (3.35) | 3.1 (3.31)
  28 Week (n=38, n=36) | 1.7 (2.61) | 2.3 (2.70)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.598, ANCOVA — P-value for treatment differences in Total score at 8 weeks; Mean Difference (Net) = -0.3, 95% CI [-1.6 to 0.9], Standard Error of Mean 0.64

9. Secondary Outcome: Nijmeegse Ouderlijke Stress Index (NOSI) Total Score
Description: The NOSI contains 123 items to be completed by the primary caregiver. Individual item scores range from 1 (completely agree) to 6 (completely disagree). Total scores range from 123 to 738.
Time Frame: Baseline, 8 weeks, 28 weeks
Population: Randomized participants with value at timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
units on a scale
  Baseline (n=42, n=44) | 368.6 (79.22) | 379.5 (78.74)
  8 Week (n=38, n=39) | 350.0 (75.07) | 368.8 (81.83)
  28 Week (n=35, n=34) | 325.2 (85.76) | 328.4 (89.23)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.318, ANCOVA — P-value for treatment differences in Total score at 8 weeks; Mean Difference (Net) = -11.2, 95% CI [-33.3 to 11.0], Standard Error of Mean 11.12

10. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Focused Attention Task - Error Rates
Description: Focused attention assessed distractibility. Child needs to identify a specific target (eg, Cherry); non-target is any other fruit. Child presses "yes" when target occurs in relevant position (eg, one of vertical positions on diamond). Child presses "no" when target is absent, or when target appears on horizontal position (irrelevant target). Error rates are percentage of missing relevant targets and percentage of false alarms in response to (irr)relevant (non)targets based on number of errors/total number of trials X 100.
Time Frame: Baseline, 8 Weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: error rate (percentage)
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
error rate (percentage)
  Irrelevant Targets Baseline (n=35, n=44) | 12.3 (13.95) | 11.8 (16.06)
  Irrelevant Targets 8 Week (n=35, n=44) | 10.0 (16.09) | 13.3 (14.36)
  Relevant Nontargets Baseline (n=35, n=44) | 5.7 (8.15) | 2.9 (5.97)
  Relevant Nontargets 8 Week (n=35, n=44) | 5.1 (9.48) | 3.3 (7.04)
  Relevant Targets Baseline (n=35, n=44) | 4.8 (5.49) | 6.9 (9.04)
  Relevant Targets 8 Week (n=35, n=44) | 7.3 (9.42) | 7.2 (14.47)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.948, Mixed Models Analysis — P-value for treatment differences in Error Rate over time; Mean Difference (Net) = -0.2, 95% CI [-5.5 to 5.2], Standard Error of Mean 2.7
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.399, Mixed Models Analysis — P-value for Treatment*Condition Error Rate irrelevant targets over time; Mean Difference (Net) = -2.9, 95% CI [-9.7 to 3.9], Standard Error of Mean 3.5
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.570, Mixed Models Analysis — P-value for Treatment*Condition Error Rate relevant nontargets over time; Mean Difference (Net) = 1.7, 95% CI [-4.3 to 7.8], Standard Deviation 3.1

11. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Focused Attention Task - Reaction Times for Hits and Correct Rejections
Description: Task is the same as described in Outcome Measure #10. Reaction times (RT) for hits are mean RTs of correct responses to relevant targets. RTs for correct rejections are mean RTs for correct rejections are mean RTs for correct no responses to irrelevant targets and relevant nontargets.
Time Frame: Baseline, 8 Weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
milliseconds
  Irrelevant Target Baseline (n=34, n=42) | 1260.1 (413.09) | 1217.3 (533.92)
  Irrelevant Target 8 Week (n=32, n=43) | 1167.8 (493.57) | 1206.0 (547.64)
  Relevant Nontarget Baseline (n=34, n=43) | 1208.4 (509.62) | 1220.9 (550.25)
  Relevant Nontarget 8 Week (n=33, n=43) | 1165.4 (570.35) | 1168.9 (569.16)
  Mean Reaction Time Hits Baseline (n=34, n=42) | 1045.6 (411.14) | 1084.4 (518.50)
  Mean Reaction Time Hits 8 Week (n=33, n=43) | 1013.0 (505.52) | 1017.7 (475.82)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.352, Mixed Models Analysis — P-value for Treatment differences in Reaction time over time; Mean Difference (Net) = -61.9, 95% CI [-193.5 to 69.8], Standard Error of Mean 66.0
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.553, Mixed Models Analysis — P-value for Treatment*Condition Mean Reaction Time correct rejections irrelevant target over time; Mean Difference (Net) = -37.1, 95% CI [-160.3 to 86.2], Standard Error of Mean 62.3
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.904, Mixed Models Analysis — P-value for Treatment*Condition Mean Reaction Time correct rejections relevant nontarget over time; Mean Difference (Net) = 7.0, 95% CI [-107.1 to 121.1], Standard Error of Mean 57.7

12. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Focused Attention Task - Standard Deviation of Reaction Times for Hits and Correct Rejections
Description: Task is the same as described in Outcome Measure #10. Standard deviations of reaction times (RT) assess intraindividual variability in RT and refer to the same conditions as those for mean reaction times described in Outcome Measure #11.
Time Frame: Baseline, 8 Weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
milliseconds
  Irrelevant Target Baseline (n=33, n=39) | 421.0 (263.84) | 429.4 (382.61)
  Irrelevant Target 8 Week (n=29, n=41) | 341.0 (259.84) | 431.7 (363.62)
  Relevant Nontarget Baseline (n=33, n=40) | 442.2 (374.99) | 565.6 (455.54)
  Relevant Nontarget 8 Week (n=30, n=41) | 442.6 (413.74) | 455.6 (376.87)
  Standard Deviation Hits Baseline (n=33, n=39) | 434.3 (302.61) | 497.9 (365.48)
  Standard Deviation Hits 8 Week (n=30, n=41) | 381.5 (286.96) | 393.9 (299.08)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.748, Mixed Models Analysis — P-value for Treatment differences in Standard Deviation of Reaction Time over time; Mean Difference (Net) = -21.3, 95% CI [-152.8 to 110.3], Standard Error of Mean 65.9
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.299, Mixed Models Analysis — P-value for Treatment*Condition Standard Deviation correct rejections irrelevant target over time; Mean Difference (Net) = -80.9, 95% CI [-234.3 to 72.5], Standard Error of Mean 77.5
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.840, Mixed Models Analysis — P-value for Treatment*Condition Standard Deviation correct rejections relevant nontarget over time; Mean Difference (Net) = 13.6, 95% CI [-119.3 to 146.5], Standard Error of Mean 67.1

13. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Memory Search Task - Error Rates
Description: The memory search task aims at measuring serial search processes to be carried out in working memory. There are 2 blocks (loads) with 40 trials each. Load 1 has 1 target to identify (e.g., an animal). A "yes" is required whenever the target is part of the displayed set of four stimuli (all animals). Load 2 has 2 targets. Whenever 1 of the targets appears in the successively displayed sets of four animals, a "yes" is required. Targets are present in 50% of trials. Error rates are the percentages of errors made in each task condition, based on the number of errors/total number of trials X 100.
Time Frame: Baseline, 8 Weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: error rate (percentage)
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
error rate (percentage)
  Absent Targets Load 2 Baseline (n=33, n=35) | 2.0 (3.52) | 4.4 (9.61)
  Absent Targets Load 2 8 Week (n=34, n=35) | 4.0 (6.83) | 4.3 (6.20)
  Absent Targets Load 1 Baseline (n=34, n=35) | 5.9 (14.06) | 5.1 (5.49)
  Absent Targets Load 1 8 Week (n=34, n=35) | 5.3 (6.96) | 7.6 (13.25)
  Present Targets Load 1 Baseline (n=34, n=35) | 6.5 (9.66) | 6.6 (6.84)
  Present Targets Load 1 8 Week (34, n=35) | 7.6 (9.07) | 7.9 (10.93)
  Present Targets Load 2 Baseline (n=33, n=35) | 9.5 (9.38) | 9.7 (10.07)
  Present Targets Load 2 8 Week (n=34, n=35) | 8.7 (10.10) | 10.1 (9.51)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis — P-value for Treatment differences in Error Rate over time; Mean Difference (Net) = 4.3, 95% CI [-1.2 to 9.9], Standard Error of Mean 2.8
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.297, Mixed Models Analysis — P-value for Treatment*Error Rate absent over time; Mean Difference (Net) = -1.8, 95% CI [-5.2 to 1.6], Standard Error of Mean 1.7
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis — P-value for Treatment*Targets Load 1 over time; Mean Difference (Net) = -5.1, 95% CI [-9.4 to -0.7], Standard Error of Mean 2.1

14. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Memory Search Task - Reaction Times for Hits and Correct Rejections
Description: Memory search task aims at measuring serial search processes to be carried out in working memory. There are 2 blocks (loads) with 40 trials each. Load 1 has 1 target to remember (one animal). A "yes" is required whenever the target is part of displayed set of 4 animals. Load 2 has 2 animals. A "yes" is required whenever one of the animals appears in successively displayed sets of 4 animals. Targets are present in 50% of the trials. Reaction time (RT) for hits is mean RT of correct "yes" responses to targets. RT correct rejections are mean RTs of correct "no" responses when target was missing.
Time Frame: Baseline, 8 Weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
milliseconds
  Load 1 Baseline (n=33, n=35) | 1051.9 (338.41) | 1010.4 (382.92)
  Load 1 8 Week (n=34, n=34) | 1014.8 (394.58) | 928.7 (301.04)
  Load 2 Baseline (n=32, n=34) | 1411.0 (357.50) | 1387.2 (595.37)
  Load 2 8 Week (n=34, n=34) | 1130.4 (460.66) | 1294.2 (552.25)
  Reaction Time Hits Load 1 Baseline (n=33, n=35) | 932.7 (295.14) | 881.7 (304.42)
  Reaction Time Hits Load 1 8 Week (n=34, n=34) | 882.4 (327.30) | 786.8 (257.19)
  Reaction Time Hits Load 2 Baseline (n=32, n=34) | 1131.5 (293.84) | 1111.8 (442.97)
  Reaction Time Hits Load 2 8 Week (n=34, n=34) | 1060.0 (343.53) | 1110.8 (445.61)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.228, Mixed Models Analysis — P-value for Treatment differences in Reaction Time over time; Mean Difference (Net) = -87.2, 95% CI [-230.4 to 56.0], Standard Error of Mean 71.7
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.260, Mixed Models Analysis — P-value for Treatment*Condition Mean Reaction Time correct rejections Load 1 over time; Mean Difference (Net) = 87.6, 95% CI [-65.6 to 240.8], Standard Error of Mean 77.3
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.239, Mixed Models Analysis — P-value for Treatment*Condition Mean Reaction Time correct rejections Load 2 over time; Mean Difference (Net) = 70.4, 95% CI [-47.3 to 188.2], Standard Error of Mean 59.5
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis — P-value for Treatment*Condition Mean Reaction Time hits Load 1 over time; Mean Difference (Net) = 122.7, 95% CI [-35.9 to 281.4], Standard Error of Mean 80.1

15. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Memory Search Task - Standard Deviation (SD) of Reaction Times for Hits and Correct Rejections
Description: Task is the same as described in Outcome Measure #14. Standard deviations of reaction times (RT) assess intraindividual variability in RT referring to the two conditions creating hits and correct rejections as mentioned in Outcome Measure #14.
Time Frame: Baseline, 8 weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
milliseconds
  Load 1 Baseline (n=32, n=35) | 406.2 (280.59) | 415.0 (324.66)
  Load 1 8 Week (n=32, n=33) | 408.2 (342.39) | 353.2 (273.16)
  Load 2 Baseline (n=31, n=34) | 515.4 (275.40) | 577.4 (340.89)
  Load 2 8 Week (n=32, n=33) | 544.9 (338.26) | 580.5 (375.88)
  SD Hits Load 1 Baseline (n=32, n=34) | 308.7 (239.10) | 320.3 (263.73)
  SD Hits Load 1 8 Week (n=33, n=33) | 261.6 (231.32) | 232.5 (165.44)
  SD Hits Load 2 Baseline (n=31, n=34) | 416.8 (226.87) | 424.6 (301.20)
  SD Hits Load 2 8 Week (n=32, n=33) | 380.6 (280.36) | 501.0 (382.32)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis — P-value for Treatment differences in Standard Deviation of Reaction Time over time; Mean Difference (Net) = -175.5, 95% CI [-351.5 to 0.5], Standard Error of Mean 88.0
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis — P-value for Treatment*Condition Standard Deviation correct rejections Load 1 over time; Mean Difference (Net) = 218.1, 95% CI [38.0 to 398.2], Standard Error of Mean 90.8
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.103, Mixed Models Analysis — P-value for Treatment*Condition Standard Deviation correct rejections Load 2 over time; Mean Difference (Net) = 173.6, 95% CI [-35.7 to 383.0], Standard Error of Mean 105.6
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis — P-value for Treatment*Condition Standard Deviation hits Load 1 over time; Mean Difference (Net) = 205.5, 95% CI [7.5 to 403.6], Standard Error of Mean 99.9

16. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Pursuit Motor Control Task - Accuracy
Description: A complex visuo-motor flexibility task that aims at measuring eye-hand co-ordination and fine motor control. By moving mouse cursor, the child is required to follow as closely as possible a target that randomly moves across the PC-screen. Accuracy is the mean distance between the mouse cursor and the moving target.
Time Frame: Baseline, 8 weeks
Population: Number of participants with baseline and non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 31 | 33
millimeters
  Baseline (n=30,n=33) | 7.8 (5.62) | 8.1 (5.49)
  8 Week (n=31,n=33) | 8.2 (6.88) | 10.1 (11.92)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis — P-value for Treatment difference in Accuracy over time; Mean Difference (Net) = -7.3, 95% CI [-16.9 to 2.3], Standard Error of Mean 4.6

17. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Pursuit Motor Control Task - Stability of Movement
Description: A complex visuo-motor flexibility task that measures eye-hand co-ordination and fine motor control. By moving mouse cursor, the child is required to follow as closely as possible a target that randomly moves across the PC-screen. Stability is within subject variability of mean distance between cursor and target.
Time Frame: Baseline, 8 weeks
Population: Number of participants with baseline and non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 31 | 33
millimeters
  Baseline (n=30,n=33) | 7.6 (8.24) | 8.2 (7.90)
  8 Week (n=31,n=33) | 8.2 (8.61) | 9.4 (9.24)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — P-value for Treatment difference in Stability of Movement over time; Mean Difference (Net) = -6.1, 95% CI [-11.2 to -1.0], Standard Error of Mean 2.4

18. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Go/No-Go Response Inhibition Task - Error Rates
Description: Measures inhibition of pre-potent responses. 24 Go signals (open squares) are presented, randomly mixed with 24 No-Go signals (closed squares). Subjects are required to press a key if a Go signal (target) appears on the screen but to withhold a response if they see a No-Go signal. Error rate is the percentage of key presses to No-Go signals/total number of trials X 100.
Time Frame: Baseline, 8 weeks
Population: Number of participants with baseline and a non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: error rate (percentage)
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 37 | 45
error rate (percentage)
  Absent Target Baseline | 8.0 (16.30) | 6.8 (8.49)
  Absent Target 8 Week | 4.5 (4.75) | 9.0 (15.07)
  Present Target Baseline | 2.0 (5.25) | 2.9 (6.14)
  Present Target 8 Week | 3.7 (10.01) | 1.9 (5.15)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.430, Mixed Models Analysis — P-value for Treatment difference in Error Rate over time; Mean Difference (Net) = 1.6, 95% CI [-2.4 to 5.7], Standard Error of Mean 2.0
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — P-value for Treatment*Condition Error Rate irrelevant targets over time; Mean Difference (Net) = -7.0, 95% CI [-11.8 to -2.2], Standard Error of Mean 2.4

19. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Flanker Interference Task - Error Rates
Description: Measures ability to neglect stimuli interfering with predefined stimulus-response coupling. Child presented with displays of 9 colored squares. Child responds to color of central square by pressing left mouse key when blue, and right mouse key when yellow. Part 1 (40 trials), surrounding squares may be same color (compatible) or different (neutral). Part 2 (80 trials), in 50% of trials, surrounding squares have color corresponding to predefined key press for other hand (incompatible). Error rates are percentages of errors in response to compatible and incompatible signals, respectively.
Time Frame: Baseline, 8 weeks
Population: Number of participants with baseline and one non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: error rate (percentages)
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 33 | 35
error rate (percentages)
  Compatible Signals Baseline (n=32, n=35) | 7.7 (9.80) | 8.5 (10.06)
  Compatible Signals 8 Week (n=33, n=35) | -2.1 (8.92) | -1.8 (11.43)
  Incompatible Signals Baseline (n=32, n=35) | 8.4 (10.33) | 9.1 (6.62)
  Incompatible Signals 8 Week (n=32, n=35) | -0.4 (11.11) | 0.1 (8.19)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.221, Mixed Models Analysis — P-value for Treatment differences in Error Rates over time; Mean Difference (Net) = -3.6, 95% CI [-9.6 to 2.3], Standard Error of Mean 2.9
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.307, Mixed Models Analysis — P-value for Treatment*Condition Error Rates compatible signals over time; Mean Difference (Net) = 2.1, 95% CI [-2.1 to 6.3], Standard Error of Mean 2.0

20. Secondary Outcome: Amsterdam Neuropsychological Tasks (ANT): Flanker Interference Task - Reaction Times
Description: Task is the same as described in Outcome Measure #19. Mean reaction times (RTs) are computed for correct responses to compatible and incompatible flankers, respectively.
Time Frame: Baseline, 8 weeks
Population: Number of participants with baseline and non-missing postbaseline value at visit.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 33 | 35
milliseconds
  Compatible Flankers Part 2 Baseline (n=31,n=34) | 863.1 (234.70) | 925.4 (384.55)
  Compatible Flankers Part 2 8 Week (n=33,n=35) | 901.1 (350.27) | 897.7 (376.63)
  Incompatible Flankers Part 2 Baseline (n=31,n=35) | 959.4 (295.32) | 976.5 (412.76)
  Incompatible Flankers Part 2 8 Week (n=33,n=35) | 931.9 (347.99) | 946.2 (419.63)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.752, Mixed Models Analysis — P-value for Treatment differences in Reaction Time over time; Mean Difference (Net) = -22.0, 95% CI [-163.1 to 119.1], Standard Error of Mean 68.9
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.564, Mixed Models Analysis — P-value for Treatment*Condition Mean Reaction Time correct rejections Load 2 over time; Mean Difference (Net) = 18.6, 95% CI [-47.0 to 84.3], Standard Error of Mean 31.9

21. Secondary Outcome: Cytochrome P450 2D6 Genotype
Description: Genotype characterization was used to determine participants' metabolic status.
Time Frame: baseline
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 49
participants
  Extensive Metabolizer | 28 | 28
  Intermediate Metabolizer | 13 | 15
  Poor Metabolizer | 6 | 6
  Missing | 1 | 0

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 39/48 | 32/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=48) | Placebo (N=49)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 14 (15) | 4 (5)
Vomiting (Gastrointestinal disorders) | 7 (10) | 5 (6)
Fatigue (General disorders) | 11 (12) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 12 (17) | 9 (13)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 4 (4)
Aggression (Psychiatric disorders) | 2 (2) | 3 (3)
Early morning awakening (Psychiatric disorders) | 5 (5) | 0 (0)
Initial insomnia (Psychiatric disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days